CLINICAL TRIAL: NCT05955313
Title: Effectiveness of Low-doses of Naltrexone (LDN) on Pain Perception and Quality of Life in Women With Vulvodynia
Brief Title: Effectiveness of Low-dose Naltrexone in Patients With Different Types of Vulvodynia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VN21
Record Dates: First submitted 2023-06-06; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Vulvodynia; Naltrexone; Quality of Life
Keywords: vulvodynia; low dose naltrexone; quality of life
MeSH Terms: conditions — Vulvodynia | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone (Experimental): NALTREXONE HYDROCHLORIDE 4,5 mg, coated oral tablets, 1xd. for 4 months
  Interventions: Drug: Naltrexone Hydrochloride
- Placebo (Placebo Comparator): Placebo, coated oral tablets, 1xd.
  Interventions: Drug: Naltrexone Hydrochloride

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — treatment of vulvodynia
  Other Names: naltrexone

SUMMARY:
Vulvodynia (Vd) is chronic functional vulvar pain, with prevalence of 3-16% and unclear etiopathology. Although Vd significantly deteriorates quality of life, the problem is marginalized, no pharmacologic treatment standards exist. Naltrexone hydrochloride is a specific opioid antagonist with slight agonist activity. There is growing body of evidence supporting the effectiveness of low-dose naltrexone (LDN) in different types of chronic pain. The main goal of this trial is to test the effect of LDN on pain perception and quality of life in women with different types of Vd. Half of the study population receives LDN and the remaining patients take placebo, according to randomization list. This RTC is quadruplet blinded.

DETAILED DESCRIPTION:
In this Randomized Controlled Trial the effectiveness of LDN in reducing chronic pain and improvement of quality of life in women with provoked, spontaneous or mixed vulvodynia is assessed on the basis of the test results recommended according to IMMPACT protocol, compared to the placebo arm. Patients remain in the study for 6 months (4 months of treatment with LDN or placebo). There are 5 visits by a gynecologist (diagnosis of vulvodynia, inclusion and exclusion criteria, randomization), nurse, psychologist and physiotherapist: screening, randomization, control telephone visit, final visit and telephone summary visit. Pain perception and quality of life estimation is reported by the patient in e-diary, validated psychology questionnaires are fulfilled and physical examination acc. Fascial Manipulation (CFMS) L. Stecco method is performed. Tolerability of LDN therapy will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Women from the age of 18 to the menopause or to the age of 50 (on the day of inclusion for testing).
2. Patients who are not pregnant and do not plan to become pregnant in the next 9 months from the inclusion in the study
3. Signing the patient's informed and voluntary consent to participate in the study.
4. General health of the patient (WHO = 0-2).
5. Diagnosis of vulvodynia.
6. Negative drug test found at the visit randomization.
7. Documented correct cytology result from 3 years ago (before the visit screening).
8. Stable dose of drugs acting on the central nervous system used min. 1 month before the screening visit and during the entire patient's participation in the study.
9. Acceptance or readiness to use a highly effective method of contraception from the screening visit throughout the study. Sexual abstinence is not accepted.
10. The ability to understand the principles of testing and operating electronic devices.

Exclusion Criteria:

1. Severe, hepatic and renal dysfunction defined as:

   i. An ASPT or ALT result 5 times the upper limit; ii. The level of bilirubin 3 times above the upper limit of normal - excluding patients with Gilbert's syndrome; iii. EGFR result below 30 ml / min / m2, on the basis of historical studies not older than 3 years before the screening visit or from the tests performed during the screening visit according with point 12 of the Protocol, version 1.0 of March 28, 2022.
2. Abuse of alcohol (more than 14 units per week) and other stimulants. 3. Taking psychoactive substances, including drugs, except for SSRI, SNRI, SARI (Trazodone), and anticonvulsants (Gabapentin, Pregabalin, Lamotrigine) in fixed doses from the screening visit.

4. Taking opioid drugs in the last 2 months before the screening visit (also in OTC preparations, eg Loperamide).

5. Taking naltrexone hydrochloride and Mysimba for weight loss at any time in your life.

6. BTA injection in the vulva in the last 4 months before the screening visit. 7. Endovascular procedures in the area of the small pelvis in the last 6 months before the screening visit.

8. Previous surgical procedures requiring general anesthesia (with general anesthesia) in the last 2 months before the screening visit.

9. Completed multidisciplinary therapeutic program in the treatment of vulvodynia in the last 4 months before the screening visit.

10. Diseases of the vulva: lichen, current contact vulvovaginitis, bacterial and / or yeast infections, other dermatological diseases, recurrent genital herpes (HSV; min 4 times / year).

11. Diagnosis of current or past serious mental disorders according to the criteria of ICD-10 and DSM-5, including psychotic and organic disorders (except depression and anxiety disorders).

12. Gynecological abnormalities requiring medical treatment: current HSIL, CIN II / III, pelvic inflammation, mixed or solid ovarian tumors, simple ovarian cysts greater than 5 cm, abnormal vaginal inter-cycle bleeding.

13. Pelvic venous diseases (PeVD), 4 criteria met on USG. 14. Pregnancy and lactation. 15. Spastic diseases: multiple sclerosis (MS), connective tissue diseases (Marfan syndrome and marfan-like syndromes), reactive arthritis (RA). 16. Vaginismus, Lamont scale 3-5 (gynecological examination impossible due to anxiety).

17. Significant and / or uncorrected disability in the field of sight or hearing, making it difficult to perform psychological tests.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness - change in pain intensity | from pre-treatment values (VISIT 2) to end of treatment values (VISIT 4) assessed for 4 months
  measured by 11-point NRS scale based on spontaneously experienced vulvar and vaginal pain and during vaginal penetration
Treatment effectiveness - change in type and severity of pain | from pre-treatment values (VISIT 2) to end of treatment values (VISIT 4) assessed for 4 months
  measured by McGill Questionnaire (SF-MPQ)
Treatment effectiveness - change in emotional functioning | from pre-treatment values (VISIT 2) to end of treatment values (VISIT 4) assessed for 4 months
  Beck Depression Inventory (BDI-II)
Patient's satisfaction | from pre-treatment values (VISIT 2) to end of treatment values (VISIT 4) assessed for 4 months
  measured by 11-point Lickert scale

SECONDARY OUTCOMES:
Treatment tolerability | throughout the treatment period (from VISIT 2 to VISIT 4) assessed for 4 months
  Assessment of the tolerability of LDN therapy based on the assessment of side effects and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Baszak-Radomańska, MD, PhD, Principal Investigator — Terpa Limited Liability Company Limited partnership
Locations (1):
- Terpa Limited Liability Company Limited Partnership, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baszak-Radomanska E, Wanczyk-Baszak J, Paszkowski T. Pilot study of testing a clinical tool for pelvic physical examination in patients with vulvodynia. Ginekol Pol. 2021 Mar 23. doi: 10.5603/GP.a2020.0168. Online ahead of print. PMID 33757151
- [Derived] Baszak-Radomanska E, Wanczyk-Baszak J, Paszkowski T. Pelvic floor examination in vulvodynia: VAMP protocol validation in correlation with central sensitization. Womens Health (Lond). 2025 Jan-Dec;21:17455057251338410. doi: 10.1177/17455057251338410. Epub 2025 Jul 1. PMID 40590401